CLINICAL TRIAL: NCT04518670
Title: Success in Comaneci-assist Coils Embolization Surveillance Study
Brief Title: Success in Comaneci-assist Coils Embolization Surveillance Study (SUCCESS)
Status: Completed | Type: Observational
Sponsor: Rapid Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-Co-001
Record Dates: First submitted 2020-08-11; First posted 2020-08-19 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-11

CONDITIONS: Intracranial Aneurysm
Keywords: Rapid Medical; aneurysm; Comaneci; Neurovascular intervention; Brain
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Comaneci Embolization Assist Device — assist in the coil embolization of wide-necked intracranial aneurysms with a neck width ≤ 10 mm.

SUMMARY:
The Comaneci Embolization Assist Device is indicated for use in the neurovasculature as a temporary endovascular device used to assist in the coil embolization of wide-necked intracranial aneurysms with a neck width ≤ 10 mm. A wide-necked intracranial aneurysm (IA) defines the neck width as ≥ 4 mm or a dome-to-neck ratio < 2.

The objective of the Postmarket Surveillance Plan is to assess safety and performance as used in postmarket clinical practice in the U.S.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a documented intracranial ruptured or unruptured aneurysm, suitable for embolization by coils.
2. Patient is considered for treatment with coil embolization assisted by the Comaneci Device for wide-necked intracranial aneurysms with neck width ≤ 10 mm. A wide-necked intracranial aneurysm is defined by the neck width as ≥ 4 mm or a dome-to-neck ratio < 2.
3. A signed informed consent by the patient or legally authorized representative

Exclusion Criteria:

1. Patient with known hypersensitivity to nickel-titanium

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Postmarket Sureveillance Study will include male or female patients with wide-necked ruptured and/or unruptured intracranial aneurysms that may require adjunctive assistance with coil embolization during the surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanel Ricardo, Dr., Principal Investigator — Baptist Neurological Institute
Locations (8):
- United States (8):
  - USA Health University Hospital, Mobile, Alabama
  - Carondelet St. Joseph's Hospital (Tenet), Tucson, Arizona
  - Santa Barbara Cottage, Santa Barbara, California
  - Los Robles, Thousand Oaks, California
  - Baptist Health Research Institute, Jacksonville, Florida
  - St. Mary's Medical Ctr (Tenet), West Palm Beach, Florida
  - University of Buffalo, Buffalo, New York
  - Texas Stroke Institute (Sarah Cannon TN), Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davies JM, Taqi MA, Coon AL, Lin LM, Bohnstedt B, Mascitelli J, Levy EI, Siddiqui A, Birnbaum L, Rodriguez P, Noufal M, Taussky P, Kilburg C, Gooch MR, Puri AS, Diaz O, Fifi JT, Majidi S, Yoo AJ, Soomro J, Bhuva P, Taylor RA, Oni-Orisan AO, Chen M, Sauvageau E, Cordina SM, Sugg RM, Singh J, Goren O, Liebeskind DS, Hanel RA. Comaneci-assisted embolization of wide-necked aneurysms: results from the SUCCESS postmarket US study. J Neurointerv Surg. 2025 Nov 19:jnis-2025-024136. doi: 10.1136/jnis-2025-024136. Online ahead of print. PMID 41260918

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated With the Comaneci: Coil embolization of wide-necked intracranial aneurysms treated with the Comaneci
Period: Overall Study
Arm/Group | Treated With the Comaneci
Started | 90
Completed | 79
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- Coil Embolization of Wide-necked Intracranial Aneurysms Treated With the Comaneci: Coil embolization of wide-necked intracranial aneurysms treated with the Comaneci
Arm/Group | Coil Embolization of Wide-necked Intracranial Aneurysms Treated With the Comaneci
Number analyzed (Participants) | 90
Age, Continuous [Mean (Full Range); unit: years] | 63 [30 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 66
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 90
Admitted with ruptured aneurysms [Count of Participants; unit: Participants] | 32
Elective cases with unruptured aneurysms. [Count of Participants; unit: Participants] | 58

OUTCOME MEASURES:

1. Primary Outcome: Periprocedural Events
Description: Rates of all adverse events occurring within 24 hours post-procedure and hospital discharge status.
Time Frame: 24 Hours post procedure
Measure: Number; unit: Events
Groups:
- Coil Embolization With Comaneci: Coil Embolization with Comaneci
Arm/Group | Coil Embolization With Comaneci
Number analyzed (Participants) | 90
Events | 79

2. Primary Outcome: Adverse Events
Description: All adverse events at discharge and up to 30 days post procedure.
Time Frame: 30 days post procedure
Measure: Number; unit: Events
Arm/Group | Coil Embolization With Comaneci
Number analyzed (Participants) | 90
Events | 150

3. Primary Outcome: Functional Status
Description: Functional status at discharge and 30 days assessed using the modified Rankin Scale (mRS).
  using the modified Rankin Scale (mRS). This scale runs from 0-6, from no symptoms to death as follows:
  * 0 - No symptoms
  * 1 - No significant disability. Able to carry out all usual activities, despite some symptoms.
  * 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  * 3 - Moderate disability. Requires some help, but able to walk unassisted.
  * 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  * 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  * 6 - Dead.
Time Frame: 30 days post procedure
Measure: Number; unit: participants
Arm/Group | Coil Embolization of Wide-necked Intracranial Aneurysms Treated With the Comaneci
Number analyzed (Participants) | 88
participants
  0 | 41
  1 | 21
  2 | 9
  3 | 5
  4 | 4
  5 | 6
  6 | 2

4. Primary Outcome: Number of Participants With Successful Intracranial Aneurysm Occlusion
Description: Successful intracranial aneurysm occlusion (measured by Raymond Roy classification I or II) at the end of procedure, using digital subtraction angiography (DSA).
Time Frame: end of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Coil Embolization of Wide-necked Intracranial Aneurysms Treated With the Comaneci
Number analyzed (Participants) | 90
Participants | 77

5. Primary Outcome: Number of Participants With Successful Intracranial Aneurysm (IA) Occlusion
Description: Successful intracranial aneurysm (IA) occlusion, that is a stable IA occlusion, measured by Raymond Roy classification I or II taken at 6 months (± 21d) post procedure without the need for re-treatment of the target IA, using DSA.
Time Frame: 6 Months Post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Coil Embolization of Wide-necked Intracranial Aneurysms Treated With the Comaneci
Number analyzed (Participants) | 75
Participants | 70

6. Primary Outcome: Number of Participants With Good Clinical Outcome
Description: Good clinical outcome- mRS shift @ 6 months (change @ 6 months from pre procedure) and tetrachotomized (0,1, 2, 3-6) mRS analysis
Time Frame: 6 Months Post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Coil Embolization of Wide-necked Intracranial Aneurysms Treated With the Comaneci
Number analyzed (Participants) | 90
Participants | 57

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Treated With the Comaneci
All-Cause Mortality (participants affected / at risk) | 4/90
Serious Adverse Events (participants affected / at risk) | 37/90
Other Adverse Events (participants affected / at risk) | 22/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated With the Comaneci (N=90)
Nervous system disorders (Nervous system disorders) | 21 (39)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2)
Cardiac disorders (Cardiac disorders) | 1 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (3)
General disorders and administration site conditions (General disorders) | 5 (5)
Infections and infestations (Infections and infestations) | 4 (5)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2)
Investigations (Investigations) | 1 (1)
Product issues (Product Issues) | 4 (4)
Psychiatric disorders (Psychiatric disorders) | 2 (2)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Vascular disorders (Vascular disorders) | 14 (16)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treated With the Comaneci (N=90)
Nervous system disorders (Nervous system disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT04518670/Prot_SAP_000.pdf